CLINICAL TRIAL: NCT04787354
Title: A Randomized Phase 3 Clinical Trial Investigating Optimal Duration of Oxaliplatin Administration in Postoperative XELOX (Oxaliplatin + Capecitabine) Adjuvant Chemotherapy for the Patients With Stage II/III Gastric Cancer
Brief Title: Optimal Duration of Oxaliplatin in Adjuvant XELOX for Gastric Cancer Patients (EXODOX)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Zang, Dae Young, Principal Investigator, Hallym University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCSG ST21-05
Record Dates: First submitted 2021-03-02; First posted 2021-03-08 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Gastric Cancer
Keywords: Stomach Neoplasms; Chemotherapy, Adjuvant; Oxaliplatin; Capecitabine
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): Standard adjuvant XELOX 8 cycles
  Oxaliplatin: 130 mg/m2/day(day 1) Capecitabine: 2,000 mg/m2/day(day 1-14), q 3weeks, total 8 cycles
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine
- Study arm (Experimental): Adjuvant XELOX 4 cycles followed by capecitabine monotherapy 4 cycles
  Oxaliplatin: 130 mg/m2/day(day 1) Capecitabine: 2,000 mg/m2/day(day 1-14), q 3weeks, 4 cycles
  followed by
  Capecitabine: 2,000 mg/m2/day(day 1-14), q 3weeks, 4 cycles
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin: 130 mg/m2/day
Drug: Capecitabine — Capecitabine: 2,000 mg/m2/day

SUMMARY:
This study aims to compare the efficacy and safety of reduced adjuvant XELOX treatment (4 cycles of XELOX followed by 4 cycles of capecitabine alone) to standard adjuvant XELOX treatment (8 cycles of XELOX).

DETAILED DESCRIPTION:
XELOX (oxaliplatin + capecitabine) combination chemotherapy is considered a standard adjuvant treatment for curatively resected gastric cancer patients after it proved its effecacy in the CLASSIC trial. Adjuvant XELOX chemotherapy is a long-term treatment with a total treatment period of 6 months and it is known that about 33% of patients cannot complete treatment schedule due to side effects. In particular, peripheral neuropathy, which is caused by the cumulative administration of oxaliplatin, is a major cause of lowering the patient's quality of life and treatment compliance, and it is known that the incidence rate increases when standard XELOX treatment is continued for more than 6 cycles. In colorectal cancer, clinical studies have been actively conducted to shorten the duration of standard adjuvant chemotherapy to reduce the peripheral sensory neuropathy caused by oxaliplatin, but there are no relevant studies in gastric cancer.

This study aims to compare the efficacy and safety of reduced adjuvant XELOX treatment (4 cycles of XELOX followed by 4 cycles of capecitabine alone) to standard adjuvant XELOX treatment (8 cycles of XELOX).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed gastric or gastroesophageal junction adenocarcinoma patients who underwent curative surgery (D1 beta or D2 resection)
* Pathologically confirmed stage II, III patients (AJCC 8th edition)
* Age 19 years and older
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 2
* Adequate marrow function (ANC > 1,500/uL, Platelet >100,000/uL, Hb > 8.0 g/dL, patients with chronic anemia who require intermittent blood transfusions can also participate in the study)
* Adequate renal function, with serum creatinine < 1.5 x upper limit of normal (ULN).
* Adequate hepatic function with serum total bilirubin ≤ 1.5 x ULN, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN
* Written, informed consent to the study

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Positive pregnancy test at baseline (postmenopausal women should be amenorrhea for at least 12 months to be considered non-fertile)
* Sexually active men and women who are not willing to implement contraception during study and until 3 months after discontinuation of study drug
* Evidence of metastasis (including cytologically confirmed malignant ascites)
* Prior systemic chemotherapy or radiation therapy for stomach cancer
* Patients who have not recovered from serious complications of gastrectomy
* History of other malignancies within the last 3 years (excluding adequately treated basal cell carcinoma of the skin, in situ cancer of the cervix, non-metastatic thyroid cancer)
* A history of clinically significant uncontrolled seizures, central nervous system disorders, or mental disorders, which make it impossible to understand the informed consent or interfere with compliance with oral drug intake
* Clinically significant (i.e., active) heart disease: e.g. unstable angina requiring medication, symptomatic coronary artery disease, congestive heart failure with NYHA grade II or higher, severe cardiac arrhythmias or acute coronary syndrome in the past 6 months (including myocardial infarction)
* Lack of integrity or malabsorption syndrome in the upper gastrointestinal tract, which is likely to affect the absorption of study drug
* Serious uncontrolled infection or other serious uncontrolled disease
* History of allograft requiring immunosuppression therapy
* Received any investigational drug or procedure within 4 weeks prior to randomization
* Active viral infection (for hepatitis B carrier, patients can be registered if HBV-DNA titer is less than 20,000 IU/mL, and are allowed to use prophylactic antiviral agents by investigator's choice)
* Active HIV infection
* Patients with peripheral sensory neuropathy with functional impairment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 976 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 3-year
  The disease-free survival (DFS) will be measured from the start of study treatment until documented tumor progression (by RECIST) or death due to any cause

SECONDARY OUTCOMES:
overall survival | 5-year
  The overall survival (OS) will be estimated from the start of study treatment until participant's death and measured using the Kaplan-Meier method
Toxicity profiles | 3-year
  Adverse events will be graded using the NCI common terminology criteria for adverse events (NCTCAE) v 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym University Medical Center, Gyeonggi-do, South Korea